CLINICAL TRIAL: NCT07079852
Title: The Acute Effects of Psilocybin on Cognition, Memory, and Brain Function
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Manoj Doss (Other)
Responsible Party: Sponsor-Investigator, Manoj Doss, Assistant Professor, University of Texas at Austin
Organization: University of Texas at Austin (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: mindflux
Record Dates: First submitted 2025-07-10; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: psilocybin; memory; cognition; psychedelics; fMRI
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: All participants will receive both interventions in counterbalanced order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled, crossover masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Capsule containing microcrystalline cellulose
  Interventions: Drug: Placebo
- psilocybin (Experimental): Capsule containing 15 mg of psilocybin
  Interventions: Drug: Psilocybin 15mg

INTERVENTIONS:
Drug: Placebo — This is an inactive control condition.
  Arms: placebo
Drug: Psilocybin 15mg — This is a moderate psychoactive dose.
  Arms: psilocybin

SUMMARY:
This study will test the effects of psilocybin on memory and cognition in healthy participants using computerized tasks and magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
In a double-blind, placebo-controlled, repeated measures design in healthy participants, this study will test the effects of psilocybin on memory and cognition in healthy individuals using computerized tasks and magnetic resonance imaging (MRI). A better understanding of the basic neurocognitive effects of psilocybin may allow for minimizing potential harms and maximizing potential benefits of psilocybin therapy.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 45-years-old.
* 3-30 lifetime psychedelic uses.
* English as a first language.
* High school education (or equivalent)
* Psychiatrically healthy (as assessed by the SCID-5).
* Medically healthy (as assessed by a physical examination and ECG).
* Willingness to attend all study sessions and complete all procedures.
* BMI between 19 and 30.

Exclusion Criteria:

* Current or past diagnosis of psychiatric disorders except panic attacks, depressive disorder, or anxiety, or disorder from ≥1 year prior.
* Current or past medical conditions that might interfere with study participation or be contraindicated for psilocybin administration (e.g., hypertension, history of stroke, cardiovascular disease, etc.)
* Current daily medications except birth control (females).
* Pregnant, nursing, or planning to become pregnant (assessed with urine pregnancy test).
* Ingestion of a psychedelic <2 months prior to an experimental session (with the exception of psilocybin administered in the context of the current study's repeated measures design).
* History of serious adverse event with a psychedelic and/or self-reported hypersensitivity to psychedelics.
* Inability to abstain from alcohol 48 hours prior to an experimental session.
* Use of other psychoactive drugs (other than caffeine or nicotine) 1 week prior to an experimental session.
* Positive urine drug screening for drugs of abuse during experimental sessions.
* Self-reported ferrous metal, metallic implants, or implanted medical devices that would preclude participation in MRI procedures, including but not limited to cochlear implants, implanted brain stimulators, and aneurysm clips.
* Self-reported past penetrating brain injury or any head injury resulting in a loss of consciousness for 30 minutes or more or post-concussive symptoms for more than seven days following a head injury.
* Self-reported claustrophobia (prohibiting MRI acquisition).
* Any other factors such as unstable housing or life-threatening circumstances, erratic behavior, etc. that are judged by the investigators to be a significant barrier to participation in the study protocol and/or to establishing rapport necessary for safe administration of psilocybin.
* Participant unwillingness to not ingest or use additional serotonergic psychedelics outside the context of study procedures for the duration of the study.
* Resting blood pressure >140/90 mm hg at study entry.
* Lifetime history of cardiomyopathy, stroke, heart disease, heart attack, tachycardia, elongated QT-interval corrected by Friderichia (> 450ms for men and > 470ms for women); clinically significant cardiac arrhythmia within 1 year of study entry; and/or abnormal electrocardiogram on study entry.
* Left-handedness (given that functional lateralizations may differ from those of right-handed individuals).

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Memory accuracy from performance on a recognition memory test | 8 weeks
  Participants will be presented with a series of pictures, and their recognition memory for these pictures will be tested by presenting pictures that they previous saw (targets) intermixed with new pictures (lures). Their task will be to respond whether a picture is "old" or "new." Hit rate = p("old"|target), False alarm rate = p("old"|lure). Memory accuracy = hit rate - false alarm rate
Neural correlates of memory as measured from fMRI | 8 weeks
  Participants will be scanned with fMRI to measure brain responses associated with memory.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin Dell Medical School, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified behavioral and fMRI data
Time Frame: Data will be available following publication of the primary findings.
Access Criteria: Anyone will be able to access the de-identified behavioral and fMRI data from Open Science Framework and OpenNeuro.

REFERENCES:
- [Background] Doss MK, Mallaroni P, Mason NL, Ramaekers JG. Psilocybin and 2C-B at Encoding Distort Episodic Familiarity. Biol Psychiatry Cogn Neurosci Neuroimaging. 2024 Oct;9(10):1048-1057. doi: 10.1016/j.bpsc.2024.06.008. Epub 2024 Jun 26. PMID 38942147
- [Background] Doss MK, Samaha J, Barrett FS, Griffiths RR, de Wit H, Gallo DA, Koen JD. Unique effects of sedatives, dissociatives, psychedelics, stimulants, and cannabinoids on episodic memory: A review and reanalysis of acute drug effects on recollection, familiarity, and metamemory. Psychol Rev. 2024 Mar;131(2):523-562. doi: 10.1037/rev0000455. Epub 2023 Dec 14. PMID 38095937